CLINICAL TRIAL: NCT03855514
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Study Of NuShield® and Standard of Care (SOC) Compared to SOC Alone For The Management Of Diabetic Foot Ulcers
Brief Title: Randomized Clinical Study Assessing NuShield Versus Standard of Care in Diabetic Foot Ulcers
Acronym: DFUs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-DFU-005-NUS
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU; Chronic Diabetic Foot Ulcer; Non-healing DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NuShield (Active Comparator): NuShield® is a sterile, dehydrated placental allograft
  Interventions: Other: NuShield
- Standard of Care (No Intervention): Standard of Care (SOC) includes, but is not limited to, surgical debridement, aggressive infection management, offloading, and maintenance of appropriate cleansing at the time of each dressing change.

INTERVENTIONS:
Other: NuShield — NuShield® is a dehydrated placental allograft.
  Arms: NuShield

SUMMARY:
This prospective, multi-center, randomized, controlled clinical study compares NuShield® plus SOC to SOC alone in subjects with chronic DFUs. NuShield® will be used along with standard of care on diabetic foot ulcers of greater than 6 weeks which have not adequately responded to conventional ulcer therapy.

DETAILED DESCRIPTION:
Two hundred (200) subjects with a chronic DFU ranging in size from 0.5cm2 and 25 cm2 will be randomized 1:1 to either NuShield® and SOC or SOC alone following the 14 day screening period. Following screening and randomization, subjects shall be seen weekly for up to 24 weeks. For subjects that heal prior to week 24, a healing confirmation visit shall occur two weeks later to confirm maintenance of complete wound closure.

Subjects that are randomized into the SOC group whose DFU has not healed by week 12 may be crossed over to receive NuShield® and followed for an additional 12-14 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old and maximum of 85 years old.
2. Subjects with a diabetic foot ulcer that is either superficial, e.g. not involving tendon, capsule, or bone; or wounds that penetrate into tendon, capsule, bone and/or joint.
3. Subjects, with the presence of Diabetes, must have a Glycosylated hemoglobin (HbA1c) ≤ 12% within 4 weeks prior to randomization
4. Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to the initial screening visit with no upper limit in duration of non-healing.
5. Subject has adequate circulation to the foot as documented by either: Skin perfusion pressure (SPP) measurement of ≥ 45 mmHg, Toe-brachial index (TBI) ≥ 0.6/ Toe pressure greater than 40, Ankle-brachial index (ABI) between 0.60 and ≤ 1.3
6. Index ulcer is a minimum of 0.5 cm2 and a maximum of 25cm2 at randomization, prior to first study treatment.
7. The index ulcer has been offloaded for 14 days prior to randomization.
8. Index ulcer has not reduced in area > 20% from Day -14 to Day 0, prior to randomization.
9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
10. Subject, or their Legally Authorized Representative (LAR), has read, understood, and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
2. Treatment with HBO wound dressings that include growth factors, bioengineered tissues, or skin substitutes within 30 days of randomization.
3. History of bone cancer or metastatic disease of the affected limb or chemotherapy within the 12 months prior to randomization.
4. Subjects with a history of more than two weeks treatment with immunosuppressants (including prednisone 10 mg daily or an equivalent does of other oral steroids cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
5. Subject is on any investigational drug(s) or therapeutic device(s) within 30 days preceding the first Screening Visit.
6. History of radiation at the ulcer site.
7. Index ulcer has been previously treated or will need to be treated with any prohibited therapies within 30 days prior to randomization.
8. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
9. Active infection at the index ulcer at the time of Randomization.
10. Acute osteomyelitis or bone infection of the affected foot, where subject has received less than 4 weeks of systemic antibiotics at the time of Screening and less than 6 weeks prior to Randomization (systemic antibiotic regimen must be completed at the time of Randomization).
11. Subject's with suspected infection who have received less than 2 weeks of systemic antibiotics, or have not had surgical resection of clinically diagnosed osteomyelitis
12. Subjects with suspected osteomyelitis who have not had an X-ray, CT scan or MRI within 14 days prior to Randomization.
13. Subject is unwilling or unable to comply with the study requirement for offloading the index wound
14. Subject is pregnant or breast feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Length of time that a wound achieves complete wound closure (CWC) | 12 weeks
  Duration (number of days) to achieve CWC from baseline to week 12 assessed between both groups

SECONDARY OUTCOMES:
Greater than 40% wound closure at week 4 from baseline | 4 weeks
  Proportion of subjects achieving ≥ 40% wound closure at Week 4 from baseline
Change in wound area | 12 weeks
  Mean percent change from baseline in wound area at Week 12
Incidence of prescribed pain and/or neuropathic medications | 12 weeks
  Cumulative amount of pain and neuropathic medications taken between baseline and Week 12 assessed between both groups.
Reduction in subject reported pain at week 12 from baseline assessed between both groups via the Numeric Pain Rating Scale (NPRS) | 12 weeks
  Mean percent change at week 12 in subject reported pain, assessed via the NPRS pain scale where 0 = no pain and 10 = worst pain imaginable, on a scale of 0 to 10.
Utilization of healthcare resources assessment | 12 weeks
  Utilization of healthcare resources through Week 12
Improvement in subject reported quality of life at week 12 from baseline assessed via the Wound-QoL (Questionnaire on quality of life with chronic wounds). | 12 weeks
  Mean percent change at week 12 from baseline in subject reported quality of life scores between both groups. The 17 item Wound-QoL tool measures the disease-specific, health-related quality of life of patients with chronic wounds. A global score is computed by averaging all 17 items where subjects answer each question on a scale of 0 to 4, where 0=not at all and 4=very much.
Time to complete wound closure (CWC) by or on 24 weeks | 24 weeks
  Length of time wounds achieve CWC at week 24 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christine McLennan, Study Director — Organogenesis Inc.
Locations (9):
- United States (9):
  - ILD Research Center, Carlsbad, California
  - Limb Preservation Platform, Fresno, California
  - University of Southern California, Los Angeles, California
  - Stanford University, Redwood City, California
  - Family Foot & Ankle Specialists, Bridgeport, Connecticut
  - Doctors Research Network, Miami, Florida
  - Extremity Healthcare, Roswell, Georgia
  - NYU Winthrop Hospital, New York, New York
  - Futuro Clinical Trials, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No